CLINICAL TRIAL: NCT02209116
Title: A RCT Comparing the Effects of Providing Clinicians and Patients With the Results of an Objective Measure of Activity and Attention (QbTest) Versus Usual Care on Diagnostic and Treatment Decision Making in Children and Young People With ADHD
Brief Title: Assessing QbTest Utility in ADHD: A Randomised Controlled Trial
Acronym: AQUA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CLAHRC-EM 14046
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: ADHD; QB Test; Activity; Attention; Children; Clinical Decision Making
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QB Open (Active Comparator): Participants and their clinician will receive results of the Qb Test
  Interventions: Other: Qb Test
- Qb Blind (Other): Participants and their clinician will be blind to the results of the Qb test
  Interventions: Other: Qb Test

INTERVENTIONS:
Other: Qb Test — Given to all participants but the results will be open or blind depending on arm allocation
  Other Names: Qb Test of Activity and Attention

SUMMARY:
Attention Deficit/Hyperactivity Disorder (ADHD)is one of the most common mental health disorders of childhood. Children with ADHD often have poor attention, are restless and hyperactive and show impulsive behaviour.

It is important to detect ADHD so young people can have access to appropriate clinical interventions.

One of the most common ways ADHD is assessed is through the clinician's opinion; however, this can vary between clinicians and is thought to be one reason why ADHD may be mis-diagnosed. Using a more objective computer tasks may help improve our understanding of ADHD. One computer task is the QbTest.

The test presents different symbols to the child, and the child has to respond by pressing a button only when a target symbol appears. The test measures the child's attention, impulsivity and movement whilst doing this task.

Although the test is thought to be a valid measure, more research needs to be conducted on this measure to see whether it helps clinicians decision making.

To see whether this test helps clinicians make a diagnosis of ADHD and helps with medication decisions, children and young people will be asked to complete the task as part of their initial assessment for ADHD. Half the participants and their clinician will have access to the QbTest result; the other half will not have access to the QbTest result until the end of the study.

Participant's parents, teachers and the clinician will also be asked to complete some questionnaires about the child's symptoms and behaviour. If the child is diagnosed with ADHD and is given medication they will be asked to complete the task again on medication. The same set of questionnaires will be completed by the parents/teachers/clinicians.

The entire sample will be followed up at 6 months and asked to complete the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-17 years (may turn 18 years during the study).
* Referred to CAMHS or community paediatrics for an ADHD assessment
* Capable of providing written informed consent (over 16)
* Parental consent (under 16)

Exclusion Criteria:

* Non-fluent English
* Suspected moderate or severe learning disability
* Previous or current diagnosis of ADHD

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 267 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of clinic appointments until correct diagnosis confirmed | By 6 months
  Number of clinic appointments until correct ADHD diagnosis is confirmed or excluded for the QBOpen (delivery of immediate QbTest feedback report) and QbBlind (delayed feedback of QbTest report) groups.

SECONDARY OUTCOMES:
Time to confirmation or exclusion of ADHD diagnosis (in days) and duration of clinic visits (in minutes). | Up to 6 months
  Time to confirmation or exclusion of ADHD diagnosis (in days) and duration of clinic visits (in minutes). This will provide supporting evidence that a reduced number of clinic visits is associated with shorter overall time to diagnosis and reduced clinic time required for assessment.

OTHER OUTCOMES:
Degree of Confidence of diagnosis | Up to 6 months
  Differences in degree of confidence of diagnosis between cases in QbOpen (QbO) and QbBlind (QbB) group. These variables will assess the utility of QbTest in aiding diagnosis (diagnostic certainty).
Stability in diagnosis and confidence between the QbO and QbB group | Up to 6 months
  Stability in diagnosis and confidence between the QbO and QbB group measured as number of patients where the primary diagnosis (ADHD confirmed or excluded) was changed at their 6 month visit to the clinic.).

CONTACTS AND LOCATIONS:
Overall Officials: Chris Hollis, MRC Psych, PhD, Principal Investigator — University of Nottingham, Nottingham HC Trust
Locations (9):
- United Kingdom (9):
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester, Greater Manchester
  - Medway NHS Foundation Trust, Gillingham, Kent
  - Bridgewater Community Healthcare NHS Trust, Wigan, Lancashire
  - Leicestershire Partnership Nhs Trust, Leicester, Leicestershire
  - United Lincolnshire Hospitals NHS Trust, Lincoln, Lincolnshire
  - Alder Hey Children's NHS Foundation Trust, Liverpool, Merseyside
  - Nottinghamshire Healthcare Nhs Trust, Nottingham, Nottinghamshire
  - Nottingham University Hospitals Nhs Trust, Nottingham, Nottinghamshire
  - Sussex Partnership NHS Foundation Trust, Worthing, Sussex

REFERENCES:
- [Background] Hall CL, Walker GM, Valentine AZ, Guo B, Kaylor-Hughes C, James M, Daley D, Sayal K, Hollis C. Protocol investigating the clinical utility of an objective measure of activity and attention (QbTest) on diagnostic and treatment decision-making in children and young people with ADHD-'Assessing QbTest Utility in ADHD' (AQUA): a randomised controlled trial. BMJ Open. 2014 Dec 1;4(12):e006838. doi: 10.1136/bmjopen-2014-006838. PMID 25448628
- [Background] Hall CL, Walker GM, Valentine AZ. Correction. Protocol investigating the clinical utility of an objective measure of activity and attention (QbTest) on diagnostic and treatment decision-making in children and young people with ADHD - 'Assessing QbTest Utility in ADHD' (AQUA): a randomised controlled trial. BMJ Open. 2015 May 6;5(5):e006838corr1. doi: 10.1136/bmjopen-2014-006838corr1. No abstract available. PMID 25948406
- [Derived] Hollis C, Hall CL, Guo B, James M, Boadu J, Groom MJ, Brown N, Kaylor-Hughes C, Moldavsky M, Valentine AZ, Walker GM, Daley D, Sayal K, Morriss R; the AQUA Trial Group. The impact of a computerised test of attention and activity (QbTest) on diagnostic decision-making in children and young people with suspected attention deficit hyperactivity disorder: single-blind randomised controlled trial. J Child Psychol Psychiatry. 2018 Dec;59(12):1298-1308. doi: 10.1111/jcpp.12921. Epub 2018 Apr 26. PMID 29700813
- [Derived] Hall CL, Valentine AZ, Walker GM, Ball HM, Cogger H, Daley D, Groom MJ, Sayal K, Hollis C. Study of user experience of an objective test (QbTest) to aid ADHD assessment and medication management: a multi-methods approach. BMC Psychiatry. 2017 Feb 10;17(1):66. doi: 10.1186/s12888-017-1222-5. PMID 28183284